CLINICAL TRIAL: NCT07239778
Title: The PEDAL Intervention - Reducing Affective Lability in Bipolar Disorder - a Randomised Controlled Trial
Brief Title: The PEDAL Intervention - Reducing Affective Lability in Bipolar Disorder
Acronym: PEDAL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Vestre Viken Hospital Trust (Other); Diakonhjemmet Hospital (Other); Lovisenberg Diakonale Hospital (Other)
Responsible Party: Principal Investigator, Trine Vik Lagerberg, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 875821; 340534 (Other Grant/Funding Number: South-East Norwegian Health Authority)
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Bipolar Disorder (BD)
Keywords: Affective lability; Bipolar disorder; Psychoeducation; Group intervention; Emotion regulation; Digital tools; eHealth
MeSH Terms: conditions — Bipolar Disorder; Emotional Regulation | interventions — MD1

STUDY DESIGN:
Masking Description: Statistical analysts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU: Traditional group psychoeducation for bipolar disorder (Active Comparator): Traditional GPP for bipolar disorder consists of 11 group sessions led by one or two trained therapists. The sessions comprise predefined topics such as the characteristics of BD, theories about etiology, managing depression and mania, psychopharmacological treatment, and lifestyle advice to enhance illness stabilization. Each session has an introductory lecture on the topic held by the therapist, small-group discussions based on the participants' experiences in this area, and plenary discussions led by the therapist. The program also provides written material for the participants to read and prepare for the relevant session, provided in a booklet. It contains the educational parts, a toolkit with a mood diary, an overview of potential "warning signs" for relapse, and an emergency plan. The toolkit is used to engage the participants in self-management of the disorder.
  Interventions: Behavioral: Traditional group psychoeducation for bipolar disorder
- PEDAL: Group psychoeducation with digital elements and focus on affective lability (Experimental): The PEDAL arm provides the 11 group sessions as described for the comparator arm, and two additional sessions that have been developed for the trial to cover topics related to affective lability and emotion regulation. Thus, in this arm there will be 13 group sessions. The format of the sessions is the same as for the TAU arm. In addition, participants in this arm will have access to an online platform with the following content: All written course material, three video tutorials for emotion regulation skills training, and an app-based mood diary that provides a dashboard where participants can monitor their mood and sleep patterns.
  Interventions: Behavioral: Group psychoeducation with digital elements and focus on affective lability

INTERVENTIONS:
Behavioral: Traditional group psychoeducation for bipolar disorder — Psychosocial intervention
  Arms: TAU: Traditional group psychoeducation for bipolar disorder
Behavioral: Group psychoeducation with digital elements and focus on affective lability — Psychosocial intervention
  Other Names: The PEDAL intervention
  Arms: PEDAL: Group psychoeducation with digital elements and focus on affective lability

SUMMARY:
PEDAL is a group-based intervention for patients with bipolar disorder that builds on the traditional group psychoeducational program (GPP) by adding digital tools and specific strategies to help manage rapid fluctuations between affective states, known as affective lability. The program's goal is to help patients learn and develop new ways to better manage their condition, with particular attention to affective lability and other difficulties with affect regulation- challenges which are not typically addressed in current treatments.

The PEDAL trial will run at five clinical sites around Oslo and Vestre Viken, aiming to recruit 120 participants with bipolar disorder. The program combines existing group sessions from GPP with new components: additional group sessions focusing on strategies for improving affect regulation such as mindfulness and distress tolerance, an online platform with all course materials including instructional videos and other resources, and an app-based mood diary. This framework maintains the benefits of regular group meetings while adding digital support tools to make the intervention more personalized and accessible.

The main aim of PEDAL is to see if the new program reduces affective lability more effectively than GPP (treatment-as-usual; TAU), and both intervention groups will be compared on the level of affective lability before and after the intervention. Several secondary outcomes like mood symptoms, suicidal thoughts, perceived stress, and quality of life will also be assessed. In terms of study design, all study sites will run the PEDAL and TAU groups in parallel, and participants will be randomly assigned to either PEDAL or TAU.

To qualify for the study, participants must be aged 18-65, diagnosed with bipolar disorder, able to participate in a group intervention, capable of providing informed consent, and have a smartphone or computer. People who have previously completed group psychoeducation, who are unable to complete the study period due to pregnancy or other factors, or those who cannot use the required technology are excluded.

In summary, PEDAL is a novel study that modernizes the existing group psychoeducational program for bipolar disorder by targeting affective lability through skills training and digital tools, while also evaluating its reception and effects in a controlled clinical trial.

DETAILED DESCRIPTION:
Bipolar disorder (BD) is a severe mental illness with significant costs for the affected individuals, their families, and society. Although a substantial proportion of individuals with BD respond relatively well to currently available treatment, sub-syndromal affective symptoms and affective lability (AL) are common and have a clear negative impact on functioning and quality of life. Targeting AL is an important new opportunity for intervention with high clinical potential through its links to severe outcomes, both independently and as a mediator of other risk factors. There is also a need for interventions that can easily be implemented in regular clinical practice. As such, we have a clear ambition of achieving efficacy and cost-efficiency, i.e., that the PEDAL intervention can be implemented in standard clinical settings without requiring substantial additional resources or structural changes. If successful, we believe that the PEDAL trial will contribute to increasing the quality and availability of treatment for patients with BD. Since group psychoeducation (GPP) is already implemented across many health regions in Norway and worldwide, there is potential for the PEDAL intervention to have both nationwide and international reach and impact if the current trial is successful.

PEDAL (PsychoEducation with Digital elements and focus on Affective Lability) is a group intervention for individuals with BD with educational and therapeutic elements. Its main purpose is to facilitate a learning and developmental process for the patient, in order to enable better self-management of the disorder. PEDAL builds on the well-established GPP program for BD, which has been found to be effective in reducing relapses and hospitalisations. GPP is likely to have further untapped potential in targeting additional burdensome aspects of BD and augmenting the didactic elements. In PEDAL, we reinforce traditional GPP through digital tools and several components targeting affective lability. In a randomised controlled trial, we will investigate whether the PEDAL intervention is superior to traditional GPP in reducing affective lability in BD. Five catchment-area-based clinical sites in and close to Oslo will participate, covering a total population of approximately 740.000. We aim to recruit 120 patients with BD to the trial.

AL is defined as rapid, excessive, and unpredictable shifts in affective states, is common in individuals with BD and adds to the illness burden. It is, however, not targeted successfully in current pharmacological or non-pharmacological treatments. Although a substantial proportion of individuals with BD respond relatively well to currently available treatment, sub-syndromal affective symptoms and AL have a clear negative impact on functioning and quality of life. Targeting AL is an important new opportunity for intervention with high clinical potential through its links to severe outcomes, both independently and as a mediator between e.g. early traumatic experiences and clinical expressions of BD.

New digital tools are promising for enhancing treatments and empowering individuals with mental disorders including BD. Such tools are increasingly used to expand mental health services' availability, flexibility, and personalization. These tools often require limited resources and enable the provision of quality health care irrespective of geographical location. Digital interventions currently in use in the mental health field include online and app-based cognitive behavioural therapy interventions, training of coping skills, and self-help programs with or without therapist guidance. The functional possibilities of digital tools align well with the objectives of psychoeducation, and such tools are increasingly used to enhance its availability and improve the personalization of delivery. So far, studies of digital interventions have not shown the anticipated effects in reducing affective episodes or hospitalisations in BD, or the effects, if present, have not been maintained at follow-up. One possible explanation could be that these interventions do not encompass interactive group sessions. Although they are still based on the principles of psychoeducation, they have omitted the group format, which is highly significant. Consequently, combining the well-established group format with digital tools directed at self-monitoring and self-management, such as an app-based mood diary and skills training sessions, may be a novel and more effective way of increasing empowerment, awareness, and engagement with the intervention.

Traditional GPP consists of modules, where predefined topics are addressed in group sessions and in paper-based written material for the participants to read and prepare for the relevant session. The most frequently used version of GPP in Norway comprises 10-12 weekly group sessions that are relatively independent of each other. The sessions cover topics such as the characteristics of BD, theories about etiology, managing depression and mania, psychopharmacological treatment and lifestyle advice to enhance illness stabilization. Each session has an introductory lecture on the topic held by the therapist, small-group discussions based on the participants' experiences in this area, and plenary discussions led by the therapist. The written material is provided in a booklet. It contains the educational parts, a toolkit with a mood diary, an overview of potential "warning signs" for relapse and an emergency plan. The toolkit is used to engage the participants in self-management of their disorder. Traditional GPP is generic in that it addresses the "standard bipolar patient", i.e. provides limited optional material targeting the specific needs of the individual participants. Furthermore, while the existing program improves several clinical outcomes in BD, it does not specifically target AL and does not appear to affect suicidality - the most severe clinical outcome possibly mediated by AL. Consequently, there is a need to incorporate additional elements to reduce suicide risk. Targeting AL through, e.g., improving affect regulation skills has the potential to do so.

The content of the PEDAL intervention:

The intervention will include the original sessions of GPP while enhancing the program with the following elements:

1. A new group session specifically addressing AL: Characteristics, and theories about etiology, as well as an introduction to relevant coping skills such as mindfulness, affect regulation strategies and distress tolerance.
2. A practical skills training group session, where mindfulness, affect regulation and distress tolerance strategies are demonstrated by a therapist.
3. An online platform with the following content:

   * All written course material for participants, including self-management tools (overview of coping strategies, emergency plan, etc.).
   * Three video tutorials for further skills training; mindfulness, affect regulation, and distress tolerance techniques.
   * All written course material, including an intervention manual for the PEDAL therapists.
   * A brief online "Clinician's booklet" for other clinicians involved in treating the patients attending the intervention.
4. App-based mood diary ("MyPEDAL").

Aims and hypotheses: The short-term and main aim of the current study is to test whether the PEDAL intervention is more efficient in reducing AL compared to traditional GPP, which is considered TAU in the current trial. We hypothesize that enhancing the traditional GPP for BD with new elements, as planned in the PEDAL intervention, will reduce AL in individuals with BD. It is also an aim to ensure that the PEDAL intervention is well received by patients and clinicians.

The PEDAL trial is a randomised controlled trial, where patients with BD will receive either TAU or the PEDAL intervention. To test whether the PEDAL intervention is more efficient than TAU in reducing AL, we will compare the two groups on pre- and post-intervention assessments of AL (primary outcome). We will also test for group differences on other relevant outcomes with important implications for individuals affected by BD such as affective symptoms, suicidal ideation, perceived stress, and quality of life. To investigate to which degree the PEDAL intervention is well received by patients and clinicians, we will conduct structured post-study evaluations of both arms.

All the clinical units participating in the PEDAL trial normally run traditional GPP 2-3 times a year with 12-16 patients in each group. Patients are referred to GPP from other units within the secondary psychiatric services and, in some cases, from general practitioners or contract psychiatrists and psychologists. All five study sites will run one TAU arm and one PEDAL arm in parallel, and patients will be randomized to TAU or PEDAL. Thus, approximately 60 participants will receive TAU, and 60 will receive PEDAL in the trial.

Inclusion and exclusion criteria: Routine criteria for participation in GPP in adult psychiatric units are as follows and will form the basis for which patients are considered candidates for the PEDAL trial: age between 18 and 65 years, a BD diagnosis, a clinical state that is considered adequate for group participation (i.e. the patient is not in a severe depressive or manic state or has severe ongoing substance abuse) and has adequate understanding of Scandinavian language. In addition, the following inclusion criteria will apply for the current trial: Ability to give informed consent and a valid DSM-5 or ICD-10 diagnosis of bipolar I, II or NOS disorder. Exclusion criteria are: Previous participation in GPP, pregnancy in a stage preventing completion of the intervention, and not owning a smartphone or computer, and/or objecting to the use a mood diary app.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar I, II or not otherwise specified disorder
* Understands Scandinavian language
* Owns and will use smartphone as part of the intervention
* Is considered eligible for group participation by treating clinician

Exclusion Criteria:

* Previous participation in group psychoeducation for bipolar disorder
* Will move, is late in pregnancy or other situation that prevents competion of trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to follow-up 1 (week 13 in TAU and week 15 in PEDAL) on the 18 item Affective Lability Scale - short form (ALS-SF) | Baseline, week 13/15 (follow-up 1) and week 37/39 (follow-up 2)
  The Affective Lability Scale is a validated self-report instrument assessing the typical pattern and level of affective lability, from 0 (not very descriptive of me) to 3 (very descriptive of me). Change = Follow-up 1 total score minus baseline total score.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS-10) | Baseline, week 13/15 (follow-up 1) and week 37/39 (follow-up 2)
  The Perceived Stress Scale (PSS) is a validated self-report measure used to assess the degree to which a person perceives their life as stressful, unpredictable, and uncontrollable over the past month. The scale consists of 10 items rated on a 5-point Likert scale from 0 (never) to 4 (very often). Higher scores indicate higher levels of perceived stress. Change=follow-up 1 total score minus baseline total score.
Quick Inventory of Depressive Symptoms - self-report version (QIDS-SR) | Baseline, week 13/15 (follow-up 1) and week 37/39 (follow-up 2)
  The Quick Inventory of Depressive Symptoms - self-report version (QIDS-SR) is a validated self-report measure to screen for and measure the severity of depressive symptoms in the past 7 days. The scale consists of 16 items rated on a 4-point Likert scale ranging from 0 (not present) to 3 (severe), where a higher score indicates more severe depression. Change= follow-up 1 total score minus baseline total score.
The Bech-Rafelsen Mania Scale (BRMS) | Baseline, week 13/15 (follow-up 1) and week 37/39 (follow-up 2)
  The Bech-Rafelsen Mania Scale (BRMS) is an 11-item clinician-rated scale used to measure the severity of manic symptoms in patients with bipolar disorder over the past 3 days. A higher score indicates more severe symptoms, with 11 items scored from 0 (no/low level) to 4 (high level) corresponding to different levels of mania, such as mild, moderate, or severe. Change= follow-up 1 total score minus baseline total score.
Difficulties in Emotion Regulation Scale - Short Form (DERS-SF) | Baseline, week 13/15 (follow-up 1) and week 37/39 (follow-up 2)
  Difficulties in Emotion Regulation Scale - Short Form (DERS-SF) is a validated 18-item self-report questionnaire used to measure difficulties in a person's capasity to regulate their emotions. The scale consists of 18 items rated on a 5-point Likert scale from 1 (almost never) to 5 (almost always), where higher scores indicate greater difficulties with emotion regulation. Change=follow-up 1 total score minus baseline total score.
WHO-5 Well-Being Index | Baseline, week 13/15 (follow-up 1) and week 37/39 (follow-up 2)
  The WHO-5 Wellbeing Index is a short, self-report questionnaire with 5 items that measures mental well-being over the past two weeks rated on a 6-point Likert scale from 5 (all of the time) to 0 (at no time).The scores are transformed into a percentage score from 0 to 100, where a higher score indicates better well-being. Change=follow-up 1 total score minus baseline total score.
EQ-5D-5L | Baseline, week 13/15 (follow-up 1) and week 37/39 (follow-up 2)
  The EQ-5D-5L is a standardized self-report questionnaire used to measure health-related quality of life across five dimensions, each with five levels of severity. It is a widely used tool for clinical and economic evaluations, and it allows for the assessment of a patient's health status irrespective of their disease and a single index value for health status. Change=follow-up 1 index value minus baseline index value.
Suicidal ideation/behavior | Baseline, week 13/15 (follow-up 1) and week 37/39 (follow-up 2)
  Simple, structured self-report form developed by the study group.

OTHER OUTCOMES:
electronic Case Report Form (eCRF) | Baseline.
  Digital questionnaire developed by the study group which will be filled in by the participants' primary clinician. The questionnaire covers demographics, illness history, past and current suicidal behavior, past and current substance use and current treatment.

CONTACTS AND LOCATIONS:
Locations (4):
- Norway (4):
  - Vestre Viken Hospital Trust (Drammen DPS), Drammen
  - Oslo University Hospital (Nydalen DPS and Søndre Oslo DPS), Oslo
  - Diakonhjemmet Hospital (Allmennpsykiatrisk poliklinikk), Oslo
  - Lovisenberg Diaconal Hospital (Section for Group Treatment), Oslo

IPD SHARING:
Plan to Share IPD: No
Data is considered too difficult to anonymise.

REFERENCES:
- [Background] Rozental A, Kottorp A, Boettcher J, Andersson G, Carlbring P. Negative Effects of Psychological Treatments: An Exploratory Factor Analysis of the Negative Effects Questionnaire for Monitoring and Reporting Adverse and Unwanted Events. PLoS One. 2016 Jun 22;11(6):e0157503. doi: 10.1371/journal.pone.0157503. eCollection 2016. PMID 27331907
- [Background] Faurholt-Jepsen M, Frokjaer VG, Nasser A, Jorgensen NR, Kessing LV, Vinberg M. Associations between the cortisol awakening response and patient-evaluated stress and mood instability in patients with bipolar disorder: an exploratory study. Int J Bipolar Disord. 2021 Mar 1;9(1):8. doi: 10.1186/s40345-020-00214-0. PMID 33644824
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Visted E, Solbakken OA, Maeland S, Fadnes LT, Bjerrum LB, Nordhus IH, Flo-Groeneboom E. Validation of a brief version of the Difficulties in Emotion Regulation Scale (DERS-16) with an older Norwegian population. Eur J Ageing. 2023 Jun 22;20(1):26. doi: 10.1007/s10433-023-00775-w. PMID 37347324
- [Background] Miola A, Cattarinussi G, Antiga G, Caiolo S, Solmi M, Sambataro F. Difficulties in emotion regulation in bipolar disorder: A systematic review and meta-analysis. J Affect Disord. 2022 Apr 1;302:352-360. doi: 10.1016/j.jad.2022.01.102. Epub 2022 Jan 29. PMID 35093412
- [Background] Dork J, Mangan E, Burns L, Dimenstein E. Affective Instability: Impact of Fluctuating Emotions on Regulation and Psychological Well-Being. Behav Sci (Basel). 2024 Sep 6;14(9):783. doi: 10.3390/bs14090783. PMID 39335997
- [Background] Rush AJ, Trivedi MH, Ibrahim HM, Carmody TJ, Arnow B, Klein DN, Markowitz JC, Ninan PT, Kornstein S, Manber R, Thase ME, Kocsis JH, Keller MB. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry. 2003 Sep 1;54(5):573-83. doi: 10.1016/s0006-3223(02)01866-8. PMID 12946886
- [Background] Lagerberg TV, Aminoff SR, Aas M, Bjella T, Henry C, Leboyer M, Pedersen G, Bellivier F, Icick R, Andreassen OA, Etain B, Melle I. Alcohol use disorders are associated with increased affective lability in bipolar disorder. J Affect Disord. 2017 Jan 15;208:316-324. doi: 10.1016/j.jad.2016.09.062. Epub 2016 Oct 14. PMID 27810713
- [Background] Licht RW, Jensen J. Validation of the Bech-Rafaelsen Mania Scale using latent structure analysis. Acta Psychiatr Scand. 1997 Nov;96(5):367-72. doi: 10.1111/j.1600-0447.1997.tb09931.x. PMID 9395155
- [Background] Aas M, Pedersen G, Henry C, Bjella T, Bellivier F, Leboyer M, Kahn JP, Cohen RF, Gard S, Aminoff SR, Lagerberg TV, Andreassen OA, Melle I, Etain B. Psychometric properties of the Affective Lability Scale (54 and 18-item version) in patients with bipolar disorder, first-degree relatives, and healthy controls. J Affect Disord. 2015 Feb 1;172:375-80. doi: 10.1016/j.jad.2014.10.028. Epub 2014 Oct 23. PMID 25451440
- [Background] Grande I, Berk M, Birmaher B, Vieta E. Bipolar disorder. Lancet. 2016 Apr 9;387(10027):1561-1572. doi: 10.1016/S0140-6736(15)00241-X. Epub 2015 Sep 18. PMID 26388529
- [Background] Joas E, Backman K, Karanti A, Sparding T, Colom F, Palsson E, Landen M. Psychoeducation for bipolar disorder and risk of recurrence and hospitalization - a within-individual analysis using registry data. Psychol Med. 2020 Apr;50(6):1043-1049. doi: 10.1017/S0033291719001053. Epub 2019 May 6. PMID 31057138
- [Background] Hidalgo-Mazzei D, Reinares M, Mateu A, Nikolova VL, Bonnin CDM, Samalin L, Garcia-Estela A, Perez-Sola V, Young AH, Strejilevich S, Vieta E, Colom F. OpenSIMPLe: A real-world implementation feasibility study of a smartphone-based psychoeducation programme for bipolar disorder. J Affect Disord. 2018 Dec 1;241:436-445. doi: 10.1016/j.jad.2018.08.048. Epub 2018 Aug 14. PMID 30145515
- [Background] Depp CA, Ceglowski J, Wang VC, Yaghouti F, Mausbach BT, Thompson WK, Granholm EL. Augmenting psychoeducation with a mobile intervention for bipolar disorder: a randomized controlled trial. J Affect Disord. 2015 Mar 15;174:23-30. doi: 10.1016/j.jad.2014.10.053. Epub 2014 Nov 8. PMID 25479050
- [Background] Faurholt-Jepsen M, Lindbjerg Tonning M, Fros M, Martiny K, Tuxen N, Rosenberg N, Busk J, Winther O, Thaysen-Petersen D, Aamund KA, Tolderlund L, Bardram JE, Kessing LV. Reducing the rate of psychiatric re-admissions in bipolar disorder using smartphones-The RADMIS trial. Acta Psychiatr Scand. 2021 May;143(5):453-465. doi: 10.1111/acps.13274. Epub 2021 Jan 26. PMID 33354769
- [Background] Faurholt-Jepsen M, Frost M, Christensen EM, Bardram JE, Vinberg M, Kessing LV. The effect of smartphone-based monitoring on illness activity in bipolar disorder: the MONARCA II randomized controlled single-blinded trial. Psychol Med. 2020 Apr;50(5):838-848. doi: 10.1017/S0033291719000710. Epub 2019 Apr 4. PMID 30944054
- [Background] Torous J, Bucci S, Bell IH, Kessing LV, Faurholt-Jepsen M, Whelan P, Carvalho AF, Keshavan M, Linardon J, Firth J. The growing field of digital psychiatry: current evidence and the future of apps, social media, chatbots, and virtual reality. World Psychiatry. 2021 Oct;20(3):318-335. doi: 10.1002/wps.20883. PMID 34505369
- [Background] Ducasse D, Jaussent I, Guillaume S, Azorin JM, Bellivier F, Belzeaux R, Bougerol T, Etain B, Gard S, Henry C, Kahn JP, Leboyer M, Loftus J, Passerieux C; FondaMental Advanced Centers of Expertise in Bipolar Disorders (FACE-BD) Collaborators; Olie E, Courtet P. Affect lability predicts occurrence of suicidal ideation in bipolar patients: a two-year prospective study. Acta Psychiatr Scand. 2017 May;135(5):460-469. doi: 10.1111/acps.12710. Epub 2017 Mar 5. PMID 28260234
- [Background] Aas M, Henry C, Bellivier F, Lajnef M, Gard S, Kahn JP, Lagerberg TV, Aminoff SR, Bjella T, Leboyer M, Andreassen OA, Melle I, Etain B. Affective lability mediates the association between childhood trauma and suicide attempts, mixed episodes and co-morbid anxiety disorders in bipolar disorders. Psychol Med. 2017 Apr;47(5):902-912. doi: 10.1017/S0033291716003081. Epub 2016 Nov 29. PMID 27894372
- [Background] Hoegh MC, Melle I, Aminoff SR, Laskemoen JF, Buchmann CB, Ueland T, Lagerberg TV. Affective lability across psychosis spectrum disorders. Eur Psychiatry. 2020 May 6;63(1):e53. doi: 10.1192/j.eurpsy.2020.44. PMID 32372737
- [Background] Gershon A, Eidelman P. Inter-episode affective intensity and instability: predictors of depression and functional impairment in bipolar disorder. J Behav Ther Exp Psychiatry. 2015 Mar;46:14-8. doi: 10.1016/j.jbtep.2014.07.005. Epub 2014 Aug 7. PMID 25164093
- [Background] Henry C, Van den Bulke D, Bellivier F, Roy I, Swendsen J, M'Bailara K, Siever LJ, Leboyer M. Affective lability and affect intensity as core dimensions of bipolar disorders during euthymic period. Psychiatry Res. 2008 May 30;159(1-2):1-6. doi: 10.1016/j.psychres.2005.11.016. Epub 2008 Mar 4. PMID 18295902
- [Background] Kallestad H, Wullum E, Scott J, Stiles TC, Morken G. The long-term outcomes of an effectiveness trial of group versus individual psychoeducation for bipolar disorders. J Affect Disord. 2016 Sep 15;202:32-8. doi: 10.1016/j.jad.2016.05.043. Epub 2016 May 24. PMID 27253214
- [Background] Michalak EE, Yatham LN, Wan DD, Lam RW. Perceived quality of life in patients with bipolar disorder. Does group psychoeducation have an impact? Can J Psychiatry. 2005 Feb;50(2):95-100. doi: 10.1177/070674370505000204. PMID 15807225
- [Background] Colom F, Vieta E, Sanchez-Moreno J, Palomino-Otiniano R, Reinares M, Goikolea JM, Benabarre A, Martinez-Aran A. Group psychoeducation for stabilised bipolar disorders: 5-year outcome of a randomised clinical trial. Br J Psychiatry. 2009 Mar;194(3):260-5. doi: 10.1192/bjp.bp.107.040485. PMID 19252157
- See also: Information about the study on sponsors website — https://www.oslo-universitetssykehus.no/avdelinger/klinikk-psykisk-helse-og-avhengighet/forsknings-og-innovasjonsavdelingen-i-pha/seksjon-klinisk-psykoseforskning/prosjekt-pedal/